CLINICAL TRIAL: NCT06937190
Title: Pre-Sleep Creatine Enhances Anaerobic Power in Recreationally Active Females
Acronym: SleepCrM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, caglar soylu, Asisstant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 162593019
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Anaerobic Performance; Sports Nutrition; Exercise Recovery; Muscle Fatigue; Creatine Supplementation; Recreational Physical Activity; Female Athletes
Keywords: Creatine Monohydrate; Pre-Sleep Supplementation; Anaerobic Power; Wingate Test; Muscle Damage Markers; Creatine Kinase (CK); Lactate Dehydrogenase (LDH); Female Exercise Performance; Nutritional Ergogenic Aid; Resistance Training; Recovery Enhancement
MeSH Terms: interventions — Creatine; maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: a creatine supplementation group or a placebo group, and they remain in that group for the duration of the trial.
Masking Description: Neither the participants nor the investigators know which intervention the participant is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Monohydrate Supplementation (Experimental): Participants will receive 5 grams of creatine monohydrate powder dissolved in water, flavored with a sugar-free agent, 30 minutes before sleep each night for 7 days.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Placebo Supplementation (Placebo Comparator): Participants will receive 5 grams of a placebo powder (maltodextrin), visually identical and similarly flavored to the creatine supplement, 30 minutes before sleep each night for 7 days.
  Interventions: Dietary Supplement: Placebo (Maltodextrin)

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Participants will receive 5 grams of creatine monohydrate powder dissolved in water, flavored with a sugar-free agent, 30 minutes before sleep each night for 7 days.
  Arms: Creatine Monohydrate Supplementation
Dietary Supplement: Placebo (Maltodextrin) — Visually identical placebo (maltodextrin powder, 5 g/day), flavored with a sugar-free agent, dissolved in water and consumed 30 minutes before sleep for 7 consecutive days.
  Arms: Placebo Supplementation

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial designed to examine the effects of pre-sleep creatine monohydrate supplementation on anaerobic performance and muscle damage markers in recreationally active females. Participants will be randomly assigned to receive either 5 grams of creatine monohydrate or a placebo 30 minutes before sleep for seven consecutive days. Anaerobic performance will be assessed using the Wingate Anaerobic Test, evaluating peak and average power output and fatigue index. Blood samples will be collected before and after the supplementation period to analyze markers of muscle damage, including creatine kinase and lactate dehydrogenase. This study aims to provide insight into the efficacy of short-term, time-specific creatine supplementation for enhancing performance and recovery.

ELIGIBILITY:
Inclusion Criteria:

Female, aged 18 to 25 years

Recreationally active (engaging in structured resistance training 3-4 times per week for the past 6 months)

Regular menstrual cycles (used for scheduling purposes)

Able and willing to provide informed consent

Agreement to maintain normal diet and training routines throughout the study

Exclusion Criteria:

History of musculoskeletal injury affecting lower or upper limbs within the past 6 months

Known allergy or intolerance to creatine or maltodextrin

Use of performance-enhancing substances or supplements within the last 30 days

Use of recovery modalities such as massage, cryotherapy, or compression garments during the study period

Current use of anti-inflammatory medication

Pregnancy or breastfeeding

Inability to comply with study protocol or scheduled assessments

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Average Power Output (Watts) - 30-Second Wingate Test | Baseline and post-intervention (Day 0 and Day 7)
  Average anaerobic power output will be calculated across the 30-second Wingate cycling test.

SECONDARY OUTCOMES:
Peak Power Output (Watts) - Wingate Test | Baseline and post-intervention (Day 0 and Day 7)
  Peak power output during the initial 5 seconds of the 30-second Wingate cycling test.
Fatigue Index (%) - Wingate Test | Baseline and post-intervention (Day 0 and Day 7)
  Calculated as the percent drop in power from peak to minimum power output during the 30-second Wingate test, indicating fatigue rate.
Serum Creatine Kinase (CK) Activity | Baseline and 24 hours post Wingate Test (Day 0 and Day 8)
  Serum creatine kinase activity will be measured as a marker of muscle damage using a spectrophotometric assay.
Serum Lactate Dehydrogenase (LDH) Activity | Baseline and 24 hours post Wingate Test (Day 0 and Day 8)
  Serum lactate dehydrogenase activity will be measured as an indicator of cell membrane permeability and muscle damage using spectrophotometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Azad University, Shabestar Branch, Shabestar, East Azerbaijan Province, Iran

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy concerns and the limited scope of this study. The study involves a small sample size, and data sharing could risk participant confidentiality. Additionally, there are currently no external collaborations or repositories arranged for data sharing.